CLINICAL TRIAL: NCT02304341
Title: Development of a Modified Pediatric Early Warning Score: a French Prospective Multicentre Regional Study.
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2011_20; PHRC2011 - 19-06 (Other: Ministry of Health, France)
Record Dates: First submitted 2013-04-25; First posted 2014-12-01 (Estimated); Last update posted 2015-11-03 (Estimated); Status verified 2015-11

CONDITIONS: Critical Illness
Keywords: critical illness; disease progression; child; severity of illness index; monitoring
MeSH Terms: conditions — Critical Illness; Disease Progression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- intermediate units: Children admitted to the paediatric inpatient unit in 7 regional hospitals French

SUMMARY:
Children are admitted in intermediate units when the severity requires continuous monitoring. In France, Resources allocated to intermediate units are determined from lists of diagnoses and associated acts to additional budget. A score to assess the severity of illness may be associated with acts to develop an activity indicator easy to use. The investigators have chosen 2 scores to assess severity in intermediate cares : the Paediatric Advanced Warning Score (PAWS) and the Bedside Pediatric Early System Score (PEWS). In France, they have not been validated. The correlation between the severity of children and the associated diagnoses and acts has not been studied. The main objective of this study is to validate these 2 scores. The secondary objective is to determine a simplified activity indicator.

ELIGIBILITY:
Inclusion Criteria:

* All children admitted to the paediatric inpatient unit

Exclusion Criteria:

* parental refusal

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children admitted to the paediatric inpatient unit in 7 regional hospitals French
Sampling Method: Probability Sample
Enrollment: 3016 (Actual)
Dates: Start 2012-09; Primary Completion 2014-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Changed inPaediatric Advanced Warning Score (PAWS) | at admission and each 8 hours, up to 5 days
  Temperature, Capillary Refill Time (CRT), respiratory rate, heart rate,neurological status, oxygen saturation, respiratory distress measure at admission, each 8 hours and if deteriorations

SECONDARY OUTCOMES:
Changed in Pediatric Early Warning System score (PEWS) | at admission and each 8 hours, up to 5 days
  heart rate, systolic blood pressure, Capillary Refill Time (CRT), respiratory rate, respiratory effort,transcutaneous oxygen saturation and oxygen therapy are measured at admission, each 8 hours and if deteriorations
Transfer in pediatric intensive care (YES/NO) | at each 8 hours, up to 5 days
  this secondary outcome is evaluated when the bedPEWS and PAWS scores are collected : at admission, each 8 hours and if deterioration

CONTACTS AND LOCATIONS:
Overall Officials: Stephane LETEURTRE, MD, Principal Investigator — Lille University Hospital
Locations (7):
- France (7):
  - Centre Hospitalier Général, Arras
  - Centre hospitalier général, Boulogne-sur-Mer
  - Centre Hospitalier Général, Cambrai
  - Centre Hospitalier Général, Douai
  - Centre Hospitalier général, Dunkirk
  - Centre Hospitalier Général, Lens
  - Centre Hospitalier Général, Roubaix

REFERENCES:
- [Derived] Lampin ME, Duhamel A, Behal H, Leteurtre S, Leclerc F, Recher M. Patient Characteristics and Severity Trajectories in a Pediatric Intermediate Care Unit. Indian J Pediatr. 2025 Feb;92(2):150-156. doi: 10.1007/s12098-023-04902-4. Epub 2023 Nov 16. PMID 37971648